CLINICAL TRIAL: NCT05239533
Title: A Phase 2 Open-label Study of Nivolumab Combined With Lutetium 177-Labeled Anti-Carbonic Anhydrase IX Monoclonal Antibody Girentuximab in Patients With Clear Cell Advanced Renal Cell Carcinoma
Brief Title: Study of Nivolumab in Combination With 177Lu-girentuximab for Kidney Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21-328
Record Dates: First submitted 2022-02-07; First posted 2022-02-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Clear Cell Renal Cell Carcinoma; Kidney Cancer; Advanced Renal Cell Carcinoma
Keywords: Nivolumab; 177Lu-girentuximab; Clear Cell Renal Cell Carcinoma; Kidney Cancer; Advanced Renal Cell Carcinoma; Memorial Sloan Kettering Cancer Center; 21-328
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Nivolumab; Single Photon Emission Computed Tomography Computed Tomography

STUDY DESIGN:
Intervention Model Description: 3+3 design to establish the maximal tolerated dose (MTD)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Safety lead-in Phase: Participants with Advanced or Metastatic Clear Cell Renal Cell Carcinoma/RCC (Experimental): Participants have Advanced or Metastatic Clear Cell Renal Cell Carcinoma/RCC. The protocol will start with a safety-lead in phase using a 3+3 design to establish the maximal tolerated dose (MTD) of 177Lu-labeled-girentuximab in combination with standard-dose nivolumab. The initial starting dose of 177Lu-labeled-girentuximab is 1804 MBq/m2 which is 75% of the single agent dose established in prior studies and will proceed as shown in the schema below. Once the MTD is established, a Simon two-stage optimal design will commence. 10 patients will be enrolled in the first stage and if no responses are observed, the study will be terminated. If 1 or more responses are observed in the first 10 patients, we will extend enrollment to a total of 29 patients (19 additional patients) in the second stage.
  Interventions: Drug: 177Lu-labeled-girentuximab; Drug: Nivolumab; Diagnostic Test: 89Zr-girentuximab PET/CT; Diagnostic Test: 177Lu whole body (WB) planar and SPECT/CT scans
- Phase 2 Participants (Experimental): Participants have Advanced or Metastatic Clear Cell Renal Cell Carcinoma/RCC. If 1 or more responses are observed in the first 10 patients, we will extend enrollment to a total of 29 patients (19 additional patients) in the second stage.
  Interventions: Drug: 177Lu-labeled-girentuximab; Drug: Nivolumab; Diagnostic Test: 89Zr-girentuximab PET/CT; Diagnostic Test: 177Lu whole body (WB) planar and SPECT/CT scans

INTERVENTIONS:
Drug: 177Lu-labeled-girentuximab — The initial starting dose/Dose Level 1 of 177Lu-labeled-girentuximab is 1804 MBq/m2. if 0/3 or 1/6 DLTs, participants will be treated at Dose Level 2 177Lu-girentuximab 2405 MBq/m2. >/= 2/6 DLTs, Dose Level -1 is 177Lu-girentuximab 1353 MBq/m2
  Once the MTD is established, a Simon two-stage optimal design will commence.
Drug: Nivolumab — Nivolumab 240mg q2wk
Diagnostic Test: 89Zr-girentuximab PET/CT — All patients will undergo a 89Zr-girentuximab PET/CT scan prior to every 177Lu-girentuximab administration
Diagnostic Test: 177Lu whole body (WB) planar and SPECT/CT scans — 177Lu whole body (WB) planar and SPECT/CT scans will be performed after each administration of 177Lu-girentuximab

SUMMARY:
The purpose of this study is to see if the combination of 177Lu-girentuximab and nivolumab is a safe and effective treatment for advanced clear cell renal cell carcinoma/ccRCC that has the CAIX protein.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced unresectable or metastatic RCC with either a component of clear cell histology or carbonic anhydrase-IX (CAIX) expression by immunohistochemistry (IHC) i. Archival tumor tissue will be requested from patients who have undergone biopsy or tumor resection as part of routine clinical care prior to study participation to confirm diagnosis. Patients may undergo pre-treatment biopsy during the screening period if archival tissue is insufficient for baseline analysis.

   Tumor specimen may include nephrectomy or metastatic site specimen.
2. At least one evaluable metastatic lesion as defined by RECIST 1.1 on zirconium-89 (89Zr)-girentuximab PET/CT
3. At least one prior line of systemic therapy, including at least one prior treatment with anti PD-1 or PD-L1antibody
4. Age ≥18 years
5. KPS ≥ 70
6. Adequate performance status and adequate organ function:

   1. ANC ≥ 1500 cells/μL
   2. WBC ≥ 2500/μL
   3. Platelet count ≥100,000/μL (without transfusion within 2 weeks prior to Cycle

      1, Day 1; thrombopoietic agent use is allowed)
   4. Hemoglobin ≥9.0 g/dL (patients may be transfused or receive erythropoietic treatment to meet this criterion)
7. AST, ALT, and alkaline phosphatase ≤ 2.5 x ULN, with the following exceptions:

   1. Patients with documented liver metastases: AST and/or ALT ≤ 5 x ULN
   2. Patients with documented liver or bone metastases: alkaline phosphatase ≤ 5 x ULN
8. Serum bilirubin ≤ 2 x ULN

   a) Patients with known Gilbert disease who have serum bilirubin level ≤ 3 x ULN may be enrolled.
9. INR and aPTT ≤ 1.5 x ULN

   a) This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
10. Creatinine clearance ≥ 40mL/min, as measured by the Cockcroft-Gault formula.
11. Women of childbearing potential and men are advised to practice double-barrier contraception until a minimum of 6 months after IV 89Zr-girentuximab or177Lu-girentuximab administration. Women of childbearing potential are advised to practice double-barrier contraception until a minimum of 5 months after nivolumab.
12. Signed consent form by the participant or a legally authorized representative (LAR).

Exclusion Criteria:

1. Renal cell carcinoma with no histological evidence of any component of clear cell features. Note: Unclassified RCC with clear cell features is eligible for inclusion.
2. Prior treatment with 177Lu- girentuximab.
3. Known hypersensitivity to girentuximab or DFO (desferoxamine).
4. Exposure to murine or chimeric antibodies within the last 5 years.
5. Previous administration of any radionuclide within 10 half-lives of the same.
6. Radiotherapy for RCC within 14 days prior to Cycle 1, Day 1 except for single-fraction radiotherapy given for the indication of pain control which should be given at least 48 hours prior to C1D1.
7. Active untreated metastases to the brain >1cm or symptomatic (of any size)
8. Active untreated metastases to the spinal cord or leptomeningeal disease
9. Patients with uncontrolled pain who are not on a stable pain regimen .
10. History of steroid requirement > 10 mg daily prednisone in the past 2 years for autoimmune comorbidities.
11. Prior checkpoint inhibitor therapy discontinued due to immune related adverse events.
12. Anti-cancer therapy within 2 weeks prior to enrollment.
13. Uncontrolled hypercalcemia (≥ 1.5 mmol/L ionized calcium or Ca ≥ 12 mg/dL or corrected serum calcium ≥ ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab.
14. Malignancies other than RCC within 3 years prior to Cycle 1, Day 1, except for those with a negligible risk of metastasis or death, treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent, non-muscle-invasive urothelial carcinoma).
15. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
16. HIV infection if not well-controlled with antiretroviral therapy
17. Patients with active or chronic hepatitis B or hepatitis C infection.
18. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 3 months, unstable arrhythmias, unstable angina, or EF < 50%.
19. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
20. History of stroke or transient ischemic attack within 6 months prior to Cycle 1, Day 1.
21. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Cycle 1, Day 1.
22. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
23. Clinical signs or symptoms of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding .
24. Evidence of abdominal free air not explained by paracentesis or recent surgical procedure.
25. Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture.
26. Major surgery within 4 weeks prior to enrollment (biopsy or line placement can be performed up to 24 hours prior to enrollment).
27. Pregnant and lactating women.
28. Patients in whom nivolumab treatment is not feasible for any reason (including financial/insurance).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerated dose (MTD) of 177Lu-girentuximab | 24 (+/- 2) weeks
  To determine the maximal tolerated dose (MTD) of 177Lu-girentuximab when given in combination with nivolumab (safety lead-in)
Overall Response Rate/ORR | 24 (+/- 2) weeks
  efficacy of the combination at the MTD of 177Lu-labelled girentuximab in patients with advanced ccRCC as assessed by best ORR by 24 (+/- 2) weeks by Response Evaluation Criteria In Solid Tumors (RECIST v1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Darren Feldman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activites), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org